CLINICAL TRIAL: NCT03156036
Title: Preoperative Chemoradiotherapy With Capecitabine With or Without Temozolomide in Patients With Locally Advanced Rectal Cancer; A Prospective Randomised Phase 2 Study Stratified by MGMT (O6-methylguanine DNA Methyltransferase) Status
Brief Title: Preoperative CRT With Capecitabine ± Temozolomide in Patients With LARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yong Sang Hong, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TemoCap2
Record Dates: First submitted 2017-05-03; First posted 2017-05-17 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Advanced Rectal Cancer
Keywords: Temozolomide; Capecitabine; MGMT
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MGMT hypermethylated Cohort A (Experimental): MGMT hypermethylated Cohort A patients will be randomised into preoperative CRT with temozolomide plus capecitabine arms. (n=86)
  Interventions: Drug: Capecitabine plus temozolomide VS Capecitabine
- MGMT hypermethylated Cohort B (Active Comparator): MGMT hypermethylated B Cohort patients will be randomised into preoperative CRT with capecitabine arms. (n=86)
  Interventions: Drug: Capecitabine plus temozolomide VS Capecitabine
- MGMT unmethylated Cohort A (Active Comparator): MGMT unmethylated A patients will be randomised into preoperative CRT with temozolomide plus capecitabine arms. (n=37)
  Interventions: Drug: Capecitabine plus temozolomide VS Capecitabine
- MGMT unmethylated Cohort B (Active Comparator): MGMT unmethylated B patients will be randomised into preoperative CRT with capecitabine arms.
  (n=37)
  Interventions: Drug: Capecitabine plus temozolomide VS Capecitabine

INTERVENTIONS:
Drug: Capecitabine plus temozolomide VS Capecitabine — For each cohort of MGMT hypermethylated versus MGMT unmethylated, patients will be randomised (ratio 1:1 for each arm) into preoperative CRT with capecitabine or preoperative CRT with temozolomide plus capecitabine arms.
  Chemotherapy during preoperative chemoradiotherapy:
  Capecitabine and temozolomide will be administered during radiotherapy with drug holidays (weekend break).
  dosage: Capecitabine 825 mg/m2 twice daily, Temozolomide 75 mg/m2/day
  Other Names: Temoram; Xeloda

SUMMARY:
This is a prospective biomarker-stratified, randomised phase II study of preoperative CRT with temozolomide plus capecitabine in patients with locally advanced rectal cancer.

The primary endpoint is pathologic complete response rates defined as total regression of the primary tumor.

For each cohort of MGMT hypermethylated versus MGMT unmethylated, patients will be randomised (ratio 1:1 for each arm) into preoperative CRT with capecitabine or preoperative CRT with temozolomide plus capecitabine arms. According to the prior phase I results, MGMT hypermethylated arm is estimated as 70% of total patients and the target pathologic complete response rate was assumed as 35% in this population when treated with preoperative CRT with temozolomide and capecitabine (15% in the standard treatment arm or those with unmethylated MGMT). Investigator would like to demonstrate the superiority in terms of pathologic complete responses when treated with preoperative CRT with temozolomide plus capecitabine in patients with locally advanced rectal cancer, and to validate the predictive role of MGMT status

DETAILED DESCRIPTION:
Preoperative chemoradiation (CRT) with fluoropyrimidine (5-fluorouracil or capecitabine) is now regarded as a standard treatment option in patients with locally advanced resectable rectal cancer and pathologic response rates and tumor regression grades after preoperative CRT have been proved to be important prognostic factors for survival outcomes.

Several studies of preoperative CRT with fluoropyrimidines plus other agents, such as oxaliplatin, irinotecan, cetuximab, and bevacizumab, have been performed to improve pathologic response rates; however, they have failed to show improved results compared to those with fluoropyrimidine alone.

Thus fluoropyrimidine alone is a standard chemotherapeutic strategy in patients with locally advanced resectable rectal cancer who will be treated with preoperative CRT at present.

Temozolomide is an oral alkylating agent, and has been proved to be effective in patients with glioblastoma or high grade anaplastic glioma when administered with concurrent radiotherapy either as adjuvant or recurrent settings.

Temozolomide has been known to deplete O6-methylguanine DNA methyltransferase (MGMT), which is one of the DNA repair enzymes, and recent studies have shown that MGMT gene silencing (lower expression by immunohistochemistry or hypermethylation by methylation-specific PCR) played a predictive marker of better responses to CRT with temozolomide in patient with glioblastoma and high grade anaplastic glioma.

Silencing of MGMT by promoter hypermethylation has been known to involve colorectal carcinogenesis pathway by the association with KRAS mutation and low-CIMP (CpG island methylation phenotype), and microsatellite instability. There have been suggestions that MGMT promoter hypermethylation played a role as a predictive factor of low recurrence in colorectal cancer patients with adjuvant oral fluoropyrimidine chemotherapy after curative surgery, and also as a predictive factor for treatment response from temozolomide in patients with metastatic colorectal cancer.

Therefore, combination chemotherapy of temozolomide plus capecitabine for rectal cancer patients when treated with preoperative CRT is worthy of investigated especially in those harbouring silenced MGMT gene as following reasons;

1. the role of temozolomide has been well established,
2. MGMT gene silencing is associated with colorectal carcinogenesis and might act as a predictive biomarker; and
3. the addition of temozolomide can be synergistic during preoperative CRT with capecitabine for rectal cancer patients.

Investigator have performed a phase I study of preoperative CRT with temozolomide plus capecitabine in patient with locally advanced rectal cancer, and the results of this study has been published The recommended dose of temozolomide was determined as 75 mg/m2 once daily when combined with standard preoperative CRT with capecitabine, there was no grade 4 adverse events and the treatment was generally well tolerated. MGMT hypermethylation was found in 72% of rectal cancer patients (16/22), and the pathologic complete responses rates were 37.5% (6/16) in patient harbouring hypermethylated MGMT versus 16.7% in those with unmethylated MGMT.

On the basis of prior trial results, Investigator concluded that preoperative CRT with temozolomide plus capecitabine is well tolerated without any notable adverse event, and is worthy of investigation especially in those harbouring MGMT gene silencing.

Investigator planned a prospective, biomarker-stratified, randomised phase II study of preoperative CRT with temozolomide plus capecitabine in patients with locally advanced rectal cancer to demonstrate the addition of temozolomide in the conventional preoperative CRT might enhance the pathologic responses in those harbouring hypermethylated MGMT.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, each patient must fulfill each of the following criteria:

  1. Histologically confirmed adenocarcinoma of the rectum
  2. Tumor located within 12cm of anal verge
  3. Clinical stage of cT3-4Nany (cStage II) or cTanyN1-2 (cStage III) by rectal MRI
  4. Available tumor samples for methylation-specific PCR (MSP) to investigate MGMT hypermethylation
  5. Male or female aged over 20 years
  6. Be ambulatory and have an Eastern Cooperative Oncology Group (ECOG) performance status0-1.
  7. No prior systemic treatment (chemotherapy, immunotherapy) or radiation therapy
  8. Adequate major organ functions as following:

     Hematopoietic function: ANC 1,500/mm3, Platelet 100,000/mm3 Hepatic function: serum bilirubin 2.0 mg/dL, AST/ALT levels 2.5 x UNL Renal function: serum creatinine UNL or Cockroft creatinine clearance 50 ml/min
  9. Be willing and able to comply with the protocol for the duration of the study.
  10. Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

- Patients will be exluded from the study for any of the following reasons:

1. Histology other than adenocarcinoma or tumor arising from inflammatory bowel disease
2. Inadequate tumor sample for MGMT MSP
3. Any evidence of systemic metastasis
4. Unresected synchronous colon cancer; endoscopically resected synchronous colon cancer of pTis or pT1 is permitted
5. Subjects unable to swallow oral medication because of such as current or impending intestinal obstructions, but bypass surgery (colostomy or ileostomy) is permitted before study treatment
6. Uncontrolled or severe cardiovascular disease:

   * New York Heart Association class III or IV heart disease.
   * Unstable angina or myocardial infarction within the past 6 months.
   * History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality.
7. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
8. Other malignancy within the past 5 years except cured non-melanomatous skin cancer, carcinoma in situ of the cervix, or thyroid papillary carcinoma.
9. Organ allografts requiring immunosuppressive therapy.
10. Psychiatric disorder or uncontrolled seizure that would preclude compliance.
11. Pregnant, nursing women or patients with reproductive potential without contraception.
12. Patients receiving a concomitant treatment with drugs interacting with 5-FU such as flucytosine, phenytoin, or warfarin et al.
13. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
14. Known hypersensitivity to any of the components of the study medications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response rate(Pathologic staging and tumor regression grade.) | 6 weeks(maximum 7 weeks)
  Surgery is after the completion of CRT

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh CR, Kim JE, Lee JS, Kim SY, Kim TW, Choi J, Kim J, Park IJ, Lim SB, Park JH, Kim JH, Choi MK, Cha Y, Baek JY, Beom SH, Hong YS. Preoperative Chemoradiotherapy With Capecitabine With or Without Temozolomide in Patients With Locally Advanced Rectal Cancer: A Prospective, Randomised Phase II Study Stratified by O6-Methylguanine DNA Methyltransferase Status: KCSG-CO17-02. Clin Oncol (R Coll Radiol). 2023 Feb;35(2):e143-e152. doi: 10.1016/j.clon.2022.10.016. Epub 2022 Nov 12. PMID 36376167